CLINICAL TRIAL: NCT07070895
Title: A Prospective Decentralized Investigation of the Effect of a Cough Management Feature Inside a Wellness Application (CoughPro) in Refractory or Unexplained Chronic Cough (RCC/UCC)
Brief Title: Cough Management Wellness App for Refractory or Unexplained Chronic Cough
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hyfe Inc (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CPCoMg-001
Record Dates: First submitted 2025-06-20; First posted 2025-07-17 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Refractory Chronic Cough; Unexplained Chronic Cough; Cough Hypersensitivity
Keywords: chronic cough; hyfe; cough monitoring; coughpro; refractory chronic cough; unexplained chronic cough; digital therapeutic; DTx; software enhanced treatment; cough management; behavioural cough suppression techniques; BCST; digital health; CoughMonitor Suite; cough tracking; cough recording; cough bouts; coughing; cough hypersensitivity; urge to cough; cough-free time; Leicester Cough Questionnaire (LCQ)
MeSH Terms: conditions — Chronic Cough; Cough

STUDY DESIGN:
Intervention Model Description: Prospective, Single-Cohort Interventional Study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cough Management (Experimental): CoughPro wellness application includes a Cough Management (CM) component, which delivers short, structured behavioral lessons (based on BCST) designed to help users recognize their urge to cough and apply cough suppression strategies in real-world settings. The Cough Management wellness feature is the key area of investigation in this study.
  Interventions: Behavioral: Cough Management; Device: CoughMonitor Suite

INTERVENTIONS:
Behavioral: Cough Management — CoughPro is a smartphone wellness application that uses algorithms to detect and count coughs continuously and passively (similar to a "step counter," but for cough). CoughPro also includes a Cough Management (CM) component, which delivers short, structured behavioral lessons (based on BCST) designed to help users recognize their urge to cough and apply cough suppression strategies in real-world settings. The Cough Management wellness feature is the key area of investigation in this study.
  The novel CM program is delivered entirely through participants' devices. The application aims to help users better understand and manage their cough by coupling real-time cough detection with self-management BCST resources:
  * Reduce cough frequency (coughs per hour).
  * Reduce cough intensity (as measured by cough bouts).
  * Improve cough-related quality of life (as reported by patients and its correlation with cough-free time as measured objectively).
  Other Names: Behavioural Cough Suppression Techniques (BCST); CoughPro
Device: CoughMonitor Suite — CoughMonitor Suite's smartwatch is used in this study to continuously, automatically, and passively monitor cough frequency in a fully privacy-preserving way - no audio is recorded, stored, or synced to the cloud, and no human is in the loop.
  Other Names: Hyfe CoughMonitor Suite; Hyfe CMS

SUMMARY:
The goal of this single-cohort clinical trial is to learn whether a smartphone-based Cough Management (CM) program can reduce cough frequency and burden in adults (21-80 years) who have refractory or unexplained chronic cough. ￼

The main questions it aims to answer are:

* Does four weeks of using the CM feature in the CoughPro app lower objective cough rate (coughs per hour) compared with each participant's one-week baseline? ￼
* Does the program also lessen cough intensity (bout metrics) and improve patient-reported quality-of-life scores on the Leicester Cough Questionnaire and PGI-S?

Participants will:

* Wear a Hyfe CoughMonitor smartwatch continuously for 6 weeks (1-week baseline, 4-week intervention, 1-week follow-up), charging it nightly. ￼
* Complete science-based in-app CM lessons based on behavioral cough-suppression therapy and practice the techniques during the 4-week intervention.
* Fill out online questionnaires (LCQ and PGI-S) at baseline and at the end of Week 4.
* Join a brief exit interview, then return the smartwatch and receive a compensation voucher.

ELIGIBILITY:
Inclusion Criteria:

* Age 21 or older.
* Currently suffering from a cough that started at least 8 weeks ago that is largely unproductive (i.e., at least 50% of the time the cough produces zero mucus that needs to be spit out or swallowed).
* Normal chest X-ray or chest CT scan at some point that was prescribed specifically for their cough.
* At least one physician visit for cough with standard-of-care therapy but inadequate symptom relief.
* Stability of treatment: willing to avoid new cough treatments during study or report changes if they occur.
* Ability to comply: willing/able to wear the watch daily for the required duration of study and to complete all required questionnaires.
* Informed consent: understanding of the study procedures and agreement to comply with protocol.

Exclusion Criteria:

* Recent upper respiratory infection (past 4 weeks).
* History of hemoptysis (coughing up blood) since onset of the current cough.
* Current smoker (incl. vaping) of any substance.
* ≥10 consecutive pack-years smoking history within <10 years prior to screening.
* Diagnosed with a chronic lung condition (COPD, emphysema, lung cancer, IPF, chronic bronchitis, asthma). Note: Suspected asthma without confirmed diagnosis or benefit from asthma therapy is not an exclusion.
* Current or past head/neck cancer.
* Difficulty swallowing.
* On ACE inhibitors, such as Benzapril (Lotensin), Captopril (Capoten), Enalapril/Enalaprilat (Vasotec oral and injectable), Fosinopril (Monopril), Lisinopril (Zestril and Prinivil), Moexipril (Univasc), Perindopril (Aceon), Quinapril (Accupril), Ramipril (Altace), and Trandolapril (Mavik)
* Prior treatment for cough by a speech-language pathologist.
* Living with another individual with a frequent cough that would interfere with monitoring.
* Participation in any cough intervention study within 30 days or 5 half-lives of the intervention.
* Major scheduled surgery during the study period.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-03-27 (Actual); Primary Completion 2025-08-08 (Actual); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Change in objective cough rate (coughs/hour) | From baseline (week minus 1) to end of Week 4
  Change in objective cough rate (coughs/hours) from baseline (week minus 1) to end of Week 4, measured by the CoughMonitor smartwatch.

SECONDARY OUTCOMES:
Change in cough intensity from baseline to end of Week 4 | Fom baseline (week minus 1) to end of week 4
  Change in cough intensity from baseline to end of Week 4, including:
  1. Number of cough bouts per day.
  2. Mean number of coughs within bouts.
Change in subjective impression of cough burden | From baseline to 4 weeks after starting the intervention.
  Change in subjective impression of cough burden using the Leicester Cough Questionnaire (LCQ) from baseline to 4 weeks after starting the intervention.
  LCQ covers the following domains (19 questions total, each with a value from 0 to 7): Physical, Psychological, Social. Domain scores are a total score from items in domain/number of items in domain (range 1-7). Total LCQ score results from the addition of domain scores with higher scores meaning a better outcome.
Change in subjective impression of cough burden | From baseline to 4 weeks after starting the intervention.
  Change in subjective impression of cough burden using the Patient Global Impression of Severity Scale in Chronic Cough (PGI-S) from baseline to 4 weeks after starting the intervention.
  Scale from 0 to 5, higher scores mean a worse outcome.

OTHER OUTCOMES:
Change in cough-free time | From baseline to end of Week 4.
  Change in cough-free time or intervals between coughs, statistical changepoint moments, and day/night distribution from baseline to end of Week 4.
Usability interview | Interview on the study duration, done at the completion of 4 weeks on Cough Management intervention.
  Usability interview evaluating the ease of use and features of the CoughPro app, following the completion of this study.

CONTACTS AND LOCATIONS:
Locations (1):
- Hyfe Inc., Wilmington, Delaware, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sundholm N, Shelly S, Wright ML, Reynolds J, Slovarp L, Gillespie AI. Effect of Behavioral Cough Suppression Therapy Delivered via Telehealth. J Voice. 2025 May;39(3):851.e1-851.e5. doi: 10.1016/j.jvoice.2022.11.015. Epub 2022 Dec 20. PMID 36550001
- [Background] Chaccour C, Sanchez-Olivieri I, Siegel S, Megson G, Winthrop KL, Botella JB, de-Torres JP, Jover L, Brew J, Kafentzis G, Galvosas M, Rudd M, Small P. Validation and accuracy of the Hyfe cough monitoring system: a multicenter clinical study. Sci Rep. 2025 Jan 6;15(1):880. doi: 10.1038/s41598-025-85341-3. PMID 39762316
- [Background] Yi B, Wang S, Xu X, Yu L. Efficacy of behavioral cough suppression therapy for refractory chronic cough or unexplained chronic cough: a meta-analysis of randomized controlled trials. Ther Adv Respir Dis. 2024 Jan-Dec;18:17534666241305952. doi: 10.1177/17534666241305952. PMID 39707881
- [Background] Chamberlain Mitchell SA, Garrod R, Clark L, Douiri A, Parker SM, Ellis J, Fowler SJ, Ludlow S, Hull JH, Chung KF, Lee KK, Bellas H, Pandyan A, Birring SS. Physiotherapy, and speech and language therapy intervention for patients with refractory chronic cough: a multicentre randomised control trial. Thorax. 2017 Feb;72(2):129-136. doi: 10.1136/thoraxjnl-2016-208843. Epub 2016 Sep 28. PMID 27682331
- [Background] Slovarp LJ, Jette ME, Gillespie AI, Reynolds JE, Barkmeier-Kraemer JM. Evaluation and Management Outcomes and Burdens in Patients with Refractory Chronic Cough Referred for Behavioral Cough Suppression Therapy. Lung. 2021 Jun;199(3):263-271. doi: 10.1007/s00408-021-00442-w. Epub 2021 Apr 5. PMID 33821355
- See also: Wellness app CoughPro used in this study — https://coughpro.com/
- See also: Publications on Hyfe's cough monitoring technology — https://www.hyfe.com/publications
- See also: CoughMonitor Suite's smartwatch used in this study for objective continuous cough monitoring — https://www.hyfe.com/cough-monitor